CLINICAL TRIAL: NCT00746044
Title: Evaluation of the Ratio of Urinary Coproporphyrins I and III as a Potential Biomarker of MRP2 Function in Man
Brief Title: Measurement of MRP2 Function Using Urinary Coproporphyrins
Acronym: COVOL
Status: Completed | Type: Observational
Sponsor: University Hospital, Tours (Other)
Responsible Party: University Hospital, Tours, University Hospital, Tours
Other Study IDs: PHAO07-CLG/COVOL
Record Dates: First submitted 2008-09-01; First posted 2008-09-03 (Estimated); Last update posted 2009-05-15 (Estimated); Status verified 2009-05

CONDITIONS: Healthy Subjects
Keywords: Healthy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 24h urine DNA
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Healthy volunteers >18y, 20 male, 20 female

SUMMARY:
Human Multidrug Related Protein 2 (MRP2) excretes several drugs and could therefore modulate their elimination. Individual's MRP2 activity is under genetic control. Thus it would be very useful to get an easily measurable biomarker reflecting individual's MRP2 activity. We aimed to investigate the ratio of urinary coproporphyrins I and III (UCP(I/I+III), known to be increased in patients with mutations in MRP2/ABCC2 gene.

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* > 18 y
* Affiliated to an health insurance

Exclusion Criteria:

* Patient not able to understand or to comply to the protocol

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 40 healthy subjects > 18 y 20 male, 20 female
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2008-02; Primary Completion 2008-04 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
Urinary coproporphyrins (I/I+III)ratio | End of three 24-hours periods

SECONDARY OUTCOMES:
ABCC2 polymorphisms | At the time of entering in the study

CONTACTS AND LOCATIONS:
Overall Officials: Chantal LE GUELLEC, Study Director — CHRU TOURS
Locations (1):
- CHRU de TOURS, Tours, France